CLINICAL TRIAL: NCT00931281
Title: A Blinded, Randomized, Nonfasting, Placebo-Controlled Study in Healthy Adults to Evaluate Safety, Tolerability, and Pharmacokinetic Profiles of Multiple Ascending Doses of ABT-450 With Ritonavir
Brief Title: Study in Healthy Adults to Evaluate Pharmacokinetics, Safety and Tolerability of ABT-450 With Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Isabelle Gaultier, Scientific Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-861
Record Dates: First submitted 2009-06-05; First posted 2009-07-02 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-09

CONDITIONS: HCV Infection
Keywords: Multiple Ascending Doses
MeSH Terms: conditions — Hepatitis C | interventions — paritaprevir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ABT-450/ritonavir
  Interventions: Drug: ABT-450; Drug: ritonavir
- 2 (Placebo Comparator): Placebo for ABT-450/placebo for ritonavir
  Interventions: Drug: Placebo for ABT-450; Drug: Placebo for ritonavir

INTERVENTIONS:
Drug: ABT-450 — capsules, QD or BID, 14 days, ascending doses
  Arms: 1
Drug: ritonavir — capsules, QD or BID, 14 days, ascending doses
  Other Names: ABT-538; Norvir
  Arms: 1
Drug: Placebo for ABT-450 — capsule, QD or BID, 14 days
  Other Names: placebo
  Arms: 2
Drug: Placebo for ritonavir — capsule, QD or BID, 14 days
  Other Names: placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety and tolerability of multiple doses of an experimental hepatitis C virus (HCV) protease inhibitor with ritonavir in healthy volunteers.

DETAILED DESCRIPTION:
This is a multiple ascending dose, non-fasting, open label, randomized study.

ELIGIBILITY:
Inclusion Criteria:

* overall healthy subjects
* non-childbearing potential females included

Exclusion Criteria:

* history of significant sensitivity to any drug
* positive test for HAV IgM, HBsAg, anti-HCV Ab or anti-HIV Ab
* history of gastrointestinal issues or procedures
* history of seizures, diabetes or cancer (except basal cell carcinoma)
* clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder
* use of tobacco or nicotine-containing products within the 6-month period prior to study drug administration
* donation or loss of 550mL or more blood volume or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration
* abnormal screening laboratory results that are considered clinically significant by the investigator
* current enrollment in another clinical study
* previous enrollment in this study
* recent (6-month) history of drug/alcohol abuse that could preclude adherence to the protocol
* pregnant or breastfeeding female
* requirement for any OTC and/or prescription medication, vitamins and/or herbal supplements on a regular basis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (blood draws, pre- and post-dose) | 17 days
Safety and Tolerability (ECGs, AEs, vitals, physical exams, routine labs) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle A Gaultier, M.S., IBMH, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 18161, Waukegan, Illinois, United States